CLINICAL TRIAL: NCT00694460
Title: A Phase II, Pilot, Randomized, Open-Label, Single-Center Study to Evaluate Immunogenicity, Safety and Booster Response of 3 Full Intramuscular Doses Versus 3 Half Intramuscular Doses Versus 3 Intradermal Doses Versus 2 Intradermal Doses of PCEC Rabies Vaccine Administered Concomitantly With Japanese Encephalitis Vaccine as a Pre-Exposure Regimen in 12 to 18 Months Old Toddlers in Thailand.
Brief Title: Evalution of Immunogenicity, Safety and Booster Response of a Rabies Vaccine Administered Concomitantly With Japanese Encephalitis Vaccine in Toddlers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Novartis, Novartis Vaccines
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M49P2
Record Dates: First submitted 2008-05-30; First posted 2008-06-10 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Rabies; Japanese Encephalitis; Pre-Exposure Prophylaxis
Keywords: rabies vaccination; pre-exposure prophylaxis; rabies virus neutralizing antibody
MeSH Terms: conditions — Rabies; Encephalitis, Japanese

ARMS (5):
- 1 (Experimental)
  Interventions: Biological: Three 1 mL doses of Rabies vaccine and two JE vaccine
- 2 (Experimental)
  Interventions: Biological: Three 0.5 mL doses of Rabies vaccine and two JE vaccine
- 3 (Experimental)
  Interventions: Biological: Three 0.1mL doses of Rabies Vaccine and two JE vaccine
- 4 (Experimental)
  Interventions: Biological: Two 0.1mL doses of Rabies vaccine and two JE vaccine
- 5 (Active Comparator)
  Interventions: Biological: Two doses of JE vaccine

INTERVENTIONS:
Biological: Three 1 mL doses of Rabies vaccine and two JE vaccine — Vaccination with purified chick embryo cell rabies vaccine 1.0 mL intramuscularly on Day 0, Day 7 and Day 28 (a total of 3 doses) and Beijing 1 strain of inactivated, lyophilized Japanese Encephalitis vaccine 0.25 mL subcutaneously on Day 0 and Day 7 (a total of 2 doses)
  Arms: 1
Biological: Three 0.5 mL doses of Rabies vaccine and two JE vaccine — Vaccination with purified chick embryo cell rabies vaccine 0.5 mL intramuscularly on Day 0, Day 7 and Day 28 (a total of 3 doses) and Beijing 1 strain of inactivated, lyophilized Japanese Encephalitis vaccine 0.25 mL subcutaneously on Day 0 and Day 7 (a total of 2 doses)
  Arms: 2
Biological: Three 0.1mL doses of Rabies Vaccine and two JE vaccine — Vaccination with purified chick embryo cell rabies vaccine 0.1 mL intradermally at one site on Day 0, Day 7 and Day 28 (a total of 3 doses) and Beijing 1 strain of inactivated, lyophilized Japanese Encephalitis vaccine 0.25 mL subcutaneously on Day 0 and Day 7 (a total of 2 doses)
  Arms: 3
Biological: Two 0.1mL doses of Rabies vaccine and two JE vaccine — Vaccination with purified chick embryo cell rabies vaccine 0.1 mL intradermally at one site on Day 0 and Day 28 (a total of 2 doses) and Beijing 1 strain of inactivated, lyophilized Japanese Encephalitis vaccine 0.25 mL subcutaneously on Day 0 and Day 7 (a total of 2 doses)
  Arms: 4
Biological: Two doses of JE vaccine — Vaccination with Beijing 1 strain of inactivated, lyophilized Japanese Encephalitis vaccine 0.25 mL only subcutaneously on Day 0 and Day 7 (a total of 2 doses)
  Arms: 5

SUMMARY:
This study evaluated the safety and immunogenicity of rabies vaccine and Japanese encephalitis vaccine in toddlers. All children developed adequate immune responses. Rabies vaccination with PCECV did not interfere with the antibody response to Japanese encephalitis vaccine. The rabies vaccine PCECV and Japanese encephalitis vaccine are safe and immunogenic when administered concomitantly to toddlers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 12-18 months old toddlers if they
* are in good health at time of entry into the study
* are available for all the visits scheduled in the study
* have been granted a written informed consent, signed by their parents

Exclusion Criteria:

* a history of rabies immunization
* a history of Japanese encephalitis immunization or disease
* a significant acute or chronic infectious disease at the time of enrollment
* fever ≥ 38.0°C (axillary) or/and significant acute or chronic infection requiring antibiotic or antiviral therapy within the past 7 days before enrollment
* being under treatment with corticosteroids, immunosuppressive drugs or other specific anti-inflammatory drugs or having taken chloroquine during the two months period before enrollment
* administration of any vaccine within the past 14 days before enrollment
* known immunodeficiency or an autoimmune disease
* history of allergy to eggs, egg products
* known hypersensitivity to neomycin, tetracycline, amphotericin-B
* planned surgery during the study period
* being enrolled in any other investigational trial contemporaneously
* the family plans to leave the area of the study site before the end of study period
* history of febrile convulsions
* history of wheezing

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2002-08; Primary Completion 2004-08 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Rabies virus neutralizing antibody concentrations | 2 years

SECONDARY OUTCOMES:
Japanese encephalitis virus neutralizing antibody titers | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Tropical Medicine, Mahidol University, Bangkok, Thailand